CLINICAL TRIAL: NCT04654156
Title: Assessment of Contrast Enhancement Boost for the Direct Identification of Pulmonary Emboli in Thoracic CT Angiography
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pedro TEIXEIRA-GONDIM, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI216
Record Dates: First submitted 2020-10-06; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pathological group: Patients with pulmonary embolism on thoracic CT angiography
  Interventions: Diagnostic Test: Contrast Boost post processing technique
- Healthy group: Patients without pulmonary embolism on thoracic CT angiography
  Interventions: Diagnostic Test: Contrast Boost post processing technique

INTERVENTIONS:
Diagnostic Test: Contrast Boost post processing technique — Contrast Enhancement Boost is a post-processing technique that uses an iodine density map generated by subtracting a pre- and post-contrast CT acquisition to artificially enhance pulmonary artery enhancement.

SUMMARY:
Pulmonary embolism is a common cardiovascular disease and thoracic CT angiography is currently considered the gold standard for its non-invasive diagnosis. However, the diagnostic performance of CT angiography can be hampered by an insufficient enhancement of pulmonary arteries. Contrast Enhancement Boost (CE Boost) is a post-processing technique using an iodine density map to artificially improve pulmonary artery enhancement.

This retrospective study compares standard CT-angiography images with CE Boost images to assess the potential improvement of diagnostic performance for the detection of pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent thoracic CT angiography for suspicion of pulmonary embolism in our institution between March and June 2018

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient referred in our institution by emergency practitioners who underwent thoracic CT angiography for clinical suspicion of pulmonary embolism between March and June 2018
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Number of thrombi within each branch of the pulmonary arteries | Between March and June 2018
  The pulmonary arteries were divided into 11 zones according to their anatomical characteristics then each visible thrombus was reported in a Excel table according to the zone where it was located

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No